CLINICAL TRIAL: NCT02461264
Title: Randomized Multicenter Trial of Two Transfusion Strategies for Patient Receiving Chemotherapy for Acute Leukemia or Hematopoietic Stem Cells With Medico-economic Evaluation of Cost Minimization.
Brief Title: Transfusion Strategy in Hematological Intensive Care Unit
Acronym: 1VERSUS2CGR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-128
Record Dates: First submitted 2015-05-28; First posted 2015-06-03 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Transfusion Related Complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARM A (Active Comparator): Two packed red blood cells will be transfused in patient with anemia defined as a hemoglobin level below 8 g / dL. Clinical and biological monitoring will be carried out later each day. If the hemoglobin is <8 g / dL, two new packed red blood cells are transfused and so on.
  Interventions: Drug: Two packed red blood cells Transfusion
- ARM B (Experimental): Single red blood packed cells Transfusion will be administered in patient with anemia defined as a hemoglobin level below 8 g/dL. Clinical and biological monitoring will be carried out later each day. If the hemoglobin is <8 g / dL, a single unit is transfused and so on.
  Interventions: Drug: Single red blood packed cells Transfusion

INTERVENTIONS:
Drug: Single red blood packed cells Transfusion
  Arms: ARM B
Drug: Two packed red blood cells Transfusion
  Arms: ARM A

SUMMARY:
Patients with acute hematological disease (acute leukemia, aplastic anemia, hematopoietic stem cells autologous or allogeneic ...) and hospitalized in an intensive care unit hematology require compensation of anemia and thrombocytopenia by blood transfusions of red blood packed cells (RBP) or platelet concentrates (PC).The AFSSAPS (Agence Française de Sécurité Sanitaire des Produits de Santé) recommendations (2002) specify the need to transfuse 2 RBP in case of symptomatic anemia usually for a hemoglobin between 6 and 10 g / dL. These recommendations allow to transfuse a single RBP for very elderly patients or in cases of associated heart disease (heart failure). A recent development (2012) on post-transfusion pulmonary edema overload recommends transfusion unit by unit for high risk patients.

More recently, a Swiss team has historically compared transfusion policies in 2 139 patients with hematological malignancies. The first group received 2 RBP transfusion in case of symptomatic anemia or hemoglobin level <6 g / dL. The other group only received 1 RBP at each transfusion. In total 2212 units in 1548 transfusions were performed and the 1 RBP transfusion policy has resulted in a 25% decrease in the number of RBP used without any complication. In a prospective single-center pilot study, we showed that transfusing a single RBP was possible without increasing the side effects of anemia, without complications and allow an overall reduction in consumption of red blood cell units.

Several meta-analyzes reported in intensive care or bleeding situations that a restrictive use of transfusions significantly reduces cardiac events, bleeding, bacterial infections and mortality. The number of patient to be treated to prevent one death is 33.

The main objective is to demonstrate in a randomized trial that the restrictive strategy (transfusion of a single unit at each transfusion) is not inferior to the liberal strategy (transfusion of 2 unit at each transfusion) in terms of severe complication. Transfusion are performed in case of hemoglobin level <8g/dL.

Key secondary objectives are to reduce the number of RBP used and the cost of hospitalization with a comparison of complications/mortality in the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients with either acute leukemia patient receiving intensive chemotherapy or autologous transplantation for lymphoma, allogeneic stem cell transplantation

Exclusion Criteria:

* ischemic heart failure
* acute promyelocytic leukemia
* ALKERAN autologous conditioning (myeloma patient)
* disseminated intravascular coagulation
* hemorrhagic syndrome
* stroke
* any vital distress at diagnosis
* creatinine clearance <50 ml/min
* liver disease with ALT (alanine aminotransferase)/AST(aspartate aminotransferase) ≥2.5 ULN (upper limit of normal) (except if related to tumor)
* pregnant female
* autoimmune hemolytic anemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-06 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Number of severe complications (grade 3 or more) | up to 1 month after the last day of hospitalization
  complications are defined as: stroke, transient ischemic attack, acute coronary syndrome, heart failure, arrhythmias or conduction cardiac disease, deep vein thrombosis, pulmonary embolism, elevated troponin, transfer to intensive care unit, death from any cause, new or progressive radiographic infiltrates, infections related to transfusion.

SECONDARY OUTCOMES:
number of RBP transfused | up to 1 month after the last day of hospitalization
Incidence of bleeding | up to 1 month after the last day of hospitalization
  number of patient with bleeding grade 3 or more
Transfusion related events | up to 1 month after the last day of hospitalization
  Number of transfusion related events defined as any complication that the physician declared to be related to the transfusion (fever, infection, pulmonary edema..)
Time to erythroid recovery | up to 1 month after the last day of hospitalization
  Time from randomization to last transfusion
Quality of life | up to 1 month after the last day of hospitalization
  Functional Assessment of Cancer Therapy and QLC30
time of aplasia | up to 1 month after the last day of hospitalization
  from 1st day with neutrophils<500 to first day with neutrophils>500/mm3
Transfusion performance | up to 24 hours
  difference between hemoglobin level before and 24 hours after transfusion
transfusion in out patient | up to 1 month after the last day of hospitalization
  number of RBP transfused after leaving the unit
Failure to respect the randomisation arm | up to 1 month after the last day of hospitalization
  number of patient in arm B that received 2 RBP instead of single RBP

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Caen, France

REFERENCES:
- [Result] Shander A, Hofmann A, Ozawa S, Theusinger OM, Gombotz H, Spahn DR. Activity-based costs of blood transfusions in surgical patients at four hospitals. Transfusion. 2010 Apr;50(4):753-65. doi: 10.1111/j.1537-2995.2009.02518.x. Epub 2009 Dec 9. PMID 20003061
- [Result] Madjdpour C, Spahn DR. Allogeneic red blood cell transfusions: efficacy, risks, alternatives and indications. Br J Anaesth. 2005 Jul;95(1):33-42. doi: 10.1093/bja/aeh290. Epub 2004 Oct 14. PMID 15486006
- [Result] Wang JK, Klein HG. Red blood cell transfusion in the treatment and management of anaemia: the search for the elusive transfusion trigger. Vox Sang. 2010 Jan;98(1):2-11. doi: 10.1111/j.1423-0410.2009.01223.x. Epub 2009 Aug 4. PMID 19682346
- [Result] Ma M, Eckert K, Ralley F, Chin-Yee I. A retrospective study evaluating single-unit red blood cell transfusions in reducing allogeneic blood exposure. Transfus Med. 2005 Aug;15(4):307-12. doi: 10.1111/j.0958-7578.2005.00592.x. PMID 16101808
- [Result] Leal-Noval SR, Munoz-Gomez M, Jimenez-Sanchez M, Cayuela A, Leal-Romero M, Puppo-Moreno A, Enamorado J, Arellano-Orden V. Red blood cell transfusion in non-bleeding critically ill patients with moderate anemia: is there a benefit? Intensive Care Med. 2013 Mar;39(3):445-53. doi: 10.1007/s00134-012-2757-z. Epub 2012 Nov 27. PMID 23184038
- [Result] Watkins TC, Clark CT. Critically ill and septic patient: is red blood cell transfusion adding to the Domino Effect? J Infus Nurs. 2013 Mar-Apr;36(2):116-21. doi: 10.1097/NAN.0b013e318282a6cd. PMID 23455973
- [Result] Robitaille N, Lacroix J, Alexandrov L, Clayton L, Cortier M, Schultz KR, Bittencourt H, Duval M. Excess of veno-occlusive disease in a randomized clinical trial on a higher trigger for red blood cell transfusion after bone marrow transplantation: a canadian blood and marrow transplant group trial. Biol Blood Marrow Transplant. 2013 Mar;19(3):468-73. doi: 10.1016/j.bbmt.2012.12.002. Epub 2012 Dec 7. PMID 23220014
- [Result] Berger MD, Gerber B, Arn K, Senn O, Schanz U, Stussi G. Significant reduction of red blood cell transfusion requirements by changing from a double-unit to a single-unit transfusion policy in patients receiving intensive chemotherapy or stem cell transplantation. Haematologica. 2012 Jan;97(1):116-22. doi: 10.3324/haematol.2011.047035. Epub 2011 Sep 20. PMID 21933858
- [Result] Carson JL, Carless PA, Hebert PC. Transfusion thresholds and other strategies for guiding allogeneic red blood cell transfusion. Cochrane Database Syst Rev. 2012 Apr 18;4(4):CD002042. doi: 10.1002/14651858.CD002042.pub3. PMID 22513904
- [Result] Salpeter SR, Buckley JS, Chatterjee S. Impact of more restrictive blood transfusion strategies on clinical outcomes: a meta-analysis and systematic review. Am J Med. 2014 Feb;127(2):124-131.e3. doi: 10.1016/j.amjmed.2013.09.017. Epub 2013 Oct 7. PMID 24331453
- [Result] Mear JB, Chantepie SP, Gac AC, Bazin A and Reman O. A restrictive transfusion Strategy allow a reduction of the number of packed red blood cells: result of a pilot study; Abstract 2217; PH-AB153 Bone marrow Transplant 2014.
- [Derived] Chantepie SP, Mear JB, Briant AR, Vilque JP, Gac AC, Cheze S, Girault S, Turlure P, Marolleau JP, Lebon D, Charbonnier A, Jardin F, Lenain P, Peyro-Saint-Paul L, Abonnet V, Dutheil JJ, Chene Y, Bazin A, Reman O, Parienti JJ. Effect of single-unit transfusion in patients treated for haematological disease including acute leukemia: A multicenter randomized controlled clinical trial. Leuk Res. 2023 Jun;129:107058. doi: 10.1016/j.leukres.2023.107058. Epub 2023 Mar 18. PMID 37080000
- [Derived] Chantepie SP, Mear JB, Guittet L, Dervaux B, Marolleau JP, Jardin F, Dutheil JJ, Parienti JJ, Vilque JP, Reman O. Transfusion strategy in hematological intensive care unit: study protocol for a randomized controlled trial. Trials. 2015 Nov 23;16:533. doi: 10.1186/s13063-015-1057-7. PMID 26592377